

## **INFORMED CONSENT**

## **Study Title:**

An investigation into neuropilates on motor function in chronic stroke: a pilot randomised feasibility study

**Document creation date:** August 4<sup>th</sup> 2020

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]

## **INFORMED CONSENT FORM**

An investigation into neuropilates on motor function in stroke: A pilot randomised feasibility study.

| 1 | Jame of Patient (Block Capitals) | Date | Signatuı | -e |
|---|---|---|---|---|
| | i consent to be contacted by rescurences a | 5 part of this rescuren study. | | |
| | I consent to be contacted by researchers a | s part of this research study. | Yes □ | No □ |
| | give informed explicit consent to have my data processed as part of his research study. | | Yes □ | No 🗆 |
| | I consent to take part in this research stud-<br>of the risks, benefits and alternatives. | y having been fully informed | Yes 🗆 | No 🗆 |
| | I have been given a copy of the Informatio consent form for my records. | n Leaflet and this completed | Yes □ | No 🗆 |
| | | ve permission for researchers to look at my medical records to get ormation. I have been assured that information about me will be it private and confidential. | | No 🗆 |
| | I am aware of the potential risks, benefits | and alternatives of this study. | Yes □ | No 🗆 |
| | I understand that I don't have to take part opt out at any time. I understand that I do opting out and I understand that opting out medical care. | on't have to give a reason for | Yes 🗆 | No 🗆 |
| | I have read and understood the <b>Information Leaflet</b> about this research project. The information has been fully explained to me and I have been able to ask questions, all of which have been answered to my satisfaction. | | | No 🗆 |